CLINICAL TRIAL: NCT00877123
Title: Prospective, Randomized, Double Blind Placebo Controled Clinical Trial to Assess the Effect of Vitamin D Supplementation on Fasting Glucose and IL-10 in Arab Women With Impaired Fasting Glucose.
Brief Title: Effect of Vitamin D Supplementation on Fasting Glucose and Interleukin-10 (IL-10) in Arab Women With Impaired Fasting Glucose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clalit Health Services (Other)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Uzi Milman, Director, Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District and the Department of Family Medicine, Faculty of Medicine, Technion- Israel Institute of Technology, HAIFA, ISRAEL., Clalit Health Services
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-09-43-CTIL
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2009-10

CONDITIONS: Obesity
Keywords: fasting glucose; obesity; arab women; interleukin; diabetes; impaired fasting glucose (IFG)
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): Intervention arm: Oral vitamin D 100,000 IU once a month for three consecutive months.
  Interventions: Drug: Oral vitamin D 100,000 IU
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral vitamin D 100,000 IU — Oral vitamin D 100,000 IU once a month for three consecutive months.
  Arms: Vitamin D
Drug: Placebo — similar placebo once a month for three consecutive months
  Arms: Placebo

SUMMARY:
Obesity, and its metabolic consequences - impaired fasting glucose (IFG) and diabetes, is highly prevalent among Arab women in Israel and the Middle East. Since life style modification is difficult to achieve in this population it is important to assess whether other modifiable risk factors can be detected. There is evidence that the homeostasis of vitamin D has a significant role in the eventual development of diabetes. Previous cross sectional studies have shown that low 25 (OH) vitamin D levels are related to glucose intolerance, diabetes, insulin resistance and metabolic syndrome. The study hypothesis is that 25(OH) vitamin D deficiency is highly prevalent among Arab women with IFG and that vitamin D supplementation may improve IFG and by that reduce the risk for future overt diabetes. Additionally, obesity is associated with a low-grade inflammation of white adipose tissue (WAT) resulting from chronic activation of the innate immune system. In obesity, there is an increased production and secretion of a wide range of inflammatory molecules including interleukin-10 (IL-10), which may have systemic effects on WAT and other organs. To that end the investigators will assess the influence of vitamin D supplementation on IL-10 and hs-CRP.

DETAILED DESCRIPTION:
Eligible women will be invited by their primary care physician to participate in the study. After signing an informed consent women will be randomized to receive oral vitamin D 100,000 IU or similar placebo once a month for three consecutive months. Pertinent clinical and demographic date will be documented and relevant laboratory test will be performed by the primary care team. One month after the third dose the same data and tests will be retrieved on each woman. Compliance with the study protocol will be enhanced and confirmed by a research assistant.

Objectives:

To assess the relationship between IFG and 25(OH) vitamin D levels in overweight Arab women.

To assess whether vitamin D supplementation significantly improves IFG. To assess whether vitamin D supplementation significantly modifies IL-10 and hs-CRP.

ELIGIBILITY:
Inclusion Criteria:

* Arab women, age 40-65
* No significant handicap or disabilities in ADL
* BMI > 25 kg/m2
* IFG of 100-125 mg/dl

Exclusion Criteria:

* Diabetes Mellitus
* Other medical conditions that may have an effect on IFG (cancer, chronic renal failure, inflammatory diseases etc)
* History of vascular disease
* Regular use of medications that may affect IFG (steroids, HRT, diuretics etc)
* Hypercalcemia (albumin corrected Ca >10.3 mg/dl)
* Inability to sign an informed consent due to mental or psychiatric ailment

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
fasting glucose | 4 months
interleukin-10 level | 4 months

SECONDARY OUTCOMES:
hs-CRP level | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Naim Shehadeh, MD, Principal Investigator — Faculty of Medicine, Technion, Haifa,; Uzi Milman, MD, Principal Investigator — Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District and the Department of Family Medicine, Faculty of Medicine, Technion- Israel Institute of Technology, HAIFA, ISRAEL.; Sophia Ish-Shalom, MD, Principal Investigator — Faculty of Medicine, Technion, Haifa,; Gila Rosen, PhD, Principal Investigator — Rambam Health Care Campus; Mira Barak,, PhD, Principal Investigator — Clalit Health Services, Haifa and Western Galilee District
Locations (1):
- Clalit Health Services, Haifa and Western Galilee District, Haifa, Israel